CLINICAL TRIAL: NCT00833534
Title: Consolidation Therapy With Lenalidomide (Revlimid®) With or Without Rituximab Followed by Maintenance Therapy With Revlimid® After Autologous/Syngeneic Transplant for Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: Lenalidomide With or Without Rituximab in Treating Patients With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma Who Have Undergone Autologous or Syngeneic Stem Cell Transplant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patient enrolled on study. Did not get patients in timely fashion. All referrals for study when assessed were not eligible.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Leona A. Holmberg, Fred Hutchinson Cancer Research Center
Masking: None | Purpose: Treatment
Other Study IDs: 2150.00; P30CA015704 (NIH); FHCRC-2150.00; IR-6846; CDR0000633628 (Registry Identifier: PDQ)
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia; Lymphoma
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Lenalidomide

ARMS (2):
- Group I (consolidation phase) (Experimental): Patients receive oral lenalidomide once daily on days 1-14. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lenalidomide
- Group II (consolidation phase) (Experimental): Patients receive lenalidomide as in group I. Patients also receive rituximab IV once on the day before the start of lenalidomide and then once between days 25-30, 50-55, and 75-80 for a total of 4 doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: lenalidomide

INTERVENTIONS:
Biological: rituximab — Given IV
  Arms: Group II (consolidation phase)
Drug: lenalidomide — Given orally

SUMMARY:
RATIONALE: Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. It is not yet known whether lenalidomide is more effective with or without rituximab in treating chronic lymphocytic leukemia or small lymphocytic lymphoma.

PURPOSE: This phase II trial is studying how well lenalidomide works when given with or without rituximab in treating patients with chronic lymphocytic leukemia or small lymphocytic lymphoma who have undergone autologous or syngeneic stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of consolidation therapy comprising lenalidomide with or without rituximab followed by maintenance therapy comprising lenalidomide in patients with chronic lymphocytic leukemia or small lymphocytic lymphoma who have undergone autologous or syngeneic stem cell transplantation.

OUTLINE:

* Consolidation phase: Patients are assigned to 1 of 2 treatment groups.

  * Group I: Patients receive oral lenalidomide once daily on days 1-14. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  * Group II: Patients receive lenalidomide as in group I. Patients also receive rituximab IV once on the day before the start of lenalidomide and then once between days 25-30, 50-55, and 75-80 for a total of 4 doses in the absence of disease progression or unacceptable toxicity.
* Maintenance phase: Beginning 2 months after completion of consolidation therapy, all patients receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 18 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 28 days and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL)

  * Any stage disease
* Prior histological documentation of CD20+ CLL or SLL
* Has undergone autologous or syngeneic stem cell transplantation comprising high-dose therapy with peripheral blood stem cell rescue within the past 30-120 days

  * No progressive disease after transplantation

    * Has had stable disease or some degree of response to transplantation
* No history of CNS involvement

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Platelet count ≥ 50,000/mm³* (transfusion independent)
* ANC ≥ 1,500/mm³*
* Total bilirubin ≤ 2 mg/mL (unless due to Gilbert's disease)
* SGOT/SGPT ≤ 2.5 times upper limit of normal
* Serum creatinine ≤ 2 mg/mL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective methods of contraception for at least 28 days before, during, and for at least 28 days after completion of study therapy
* Patients and their physician must be registered in the RevAssist® program and be willing and able to comply with the requirements of RevAssist®
* LVEF ≥ 45% immediately prior to transplant
* No uncontrolled congestive heart disease
* No history of myocardial infarction or coronary artery disease
* No peripheral neuropathy ≥ grade 3
* No allergy to lenalidomide, thalidomide, allopurinol, or rituximab
* No known hepatitis B, hepatitis C, or HIV seropositivity
* No other malignancies within the past 5 years, except for adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast
* No concurrent serious uncontrolled medical or psychiatric illness, including serious infection NOTE: *For 5 calendar days after transplant

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior CD34-selected stem cell product
* No chemotherapy or biologic therapy for CLL after transplant
* Prior rituximab administered before stem cell collection allowed
* Prior lenalidomide administered before transplant allowed provided patient responded to lenalidomide
* No concurrent sargramostim (GM-CSF)
* No other concurrent anticancer therapies, including radiotherapy or thalidomide
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02

PRIMARY OUTCOMES:
Efficacy of lenalidomide with or without rituximab as consolidation therapy and lenalidomide as maintenance therapy
Disease-free survival at 2 years after transplant

SECONDARY OUTCOMES:
Toxicity during consolidation and maintenance therapy as assessed by NCI CTCAE v3.0
Ability to complete planned therapy
Complete hematological remission, including bone marrow IgH remission status as assessed by PCR after consolidation and maintenance therapy
Time to disease progression
Relapse rates

CONTACTS AND LOCATIONS:
Overall Officials: Leona A. Holmberg, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Center